CLINICAL TRIAL: NCT01922609
Title: Prediction of Carotid Occlusion Intolerance by Transcranial Doppler Evaluation in Patients Undergoing Carotid Artery Stenting With Proximal Flow Arrest Protection System.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Miloslav Spacek, MD, Miloslav Spacek, MD, University Hospital, Motol
Other Study IDs: EK-1075/13
Record Dates: First submitted 2013-08-11; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Carotid Occlusion Intolerance
Keywords: Carotid stenting; Proximal protection system; Transcranial Doppler ultrasound; Cerebrovascular reserve

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal cerebrovascular reserve: Patients without preprocedural TCD signs of impaired cerebrovascular reserve
- Impaired cerebrovascular reserve: Patients with preprocedural TCD signs of impaired cerebrovascular reserve

SUMMARY:
The aim of this observational pilot study is to determine whether intolerance of carotid occlusion during carotid artery stenting can be predicted with preprocedural transcranial Doppler evaluation.

DETAILED DESCRIPTION:
Carotid artery stenting procedures are increasingly performed with devices that involve endovascular clamping of the common carotid artery, thus exposing the ipsilateral hemisphere to hypoperfusion. Approximately 5% of patients do not tolerate the clamp and are in increased risk of periprocedural cerebrovascular complication such as transient ischemic attack or stroke. To date, there is no method available that could be used to predict the risk of occlusion intolerance. The aim of this study is to determine whether preprocedural evaluation with transcranial Doppler ultrasonography can be effective in prediction of occlusion intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Either >50% symptomatic carotid artery stenosis (transient ischemic attack or ischemic stroke within 6 months before procedure) or >70% asymptomatic carotid artery stenosis eligible for carotid artery stenting with proximal flow arrest protection
* Signed informed consent

Exclusion Criteria:

* Disagreement to be included in the study
* Inadequate acoustic window for transcranial Doppler ultrasound monitoring
* Carotid occlusion
* Significant extracranial artery stenosis (>50%) other than target artery
* Inability to hold breath for sufficient time (approximately 30s)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with carotid artery stenosis indicated for carotid artery stenting with the use of proximal flow arrest protection device.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Carotid occlusion intolerance | During carotid stenting procedure
  Intolerance of carotid occlusion during carotid artery stenting detected by means of transcranial Doppler evaluation or by clinical signs of occlusion intolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Miloslav Spacek, MD, Principal Investigator — Department of cardiology, University Hospital Motol; Josef Veselka, MD, PhD, Study Chair — Department of cardiology, University Hospital Motol
Locations (1):
- Department of Cardiology, University Hospital Motol, Prague, Czech Republic, Czechia